CLINICAL TRIAL: NCT06560905
Title: Preoperative Planning With PSMA-PET in Melanoma Surgery Trial
Acronym: PPPIMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCR5614
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: All patients will receive PSMA-PET-CT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA PET-CT (Experimental): Within the two weeks prior to surgery, the patients will undergo both PSMA PET-CT & FDG PET-CT scans at least 48 hours apart.
  The Investigational Medicinal Product (IMP) under investigation in this trial is 68Ga-PSMA. This is an imaging radionuclide tracer.
  Interventions: Drug: 68Ga-PSMA

INTERVENTIONS:
Drug: 68Ga-PSMA — This is an imaging radionuclide tracer and is in chemical form. Up to 200 MBq. Route of administration is Intravenous.

SUMMARY:
This is a non-randomised, single-centre Phase 2 study, investigating whether the diagnostic biomarker, prostate-specific membrane antigen (PSMA), can detect melanoma metastases using PSMA PET/ CT.

DETAILED DESCRIPTION:
The proposed 'Preoperative Planning PSMA-PET in Melanoma Surgery (PPPIMS)' trial is a Phase 2 study, investigating the ability of PSMA as a biomarker to accurately detect melanoma metastases in patients with palpable lymphadenopathy and oligometastatic melanoma. If proven to have diagnostic utility, it may allow more precise 3D lymphatic mapping and identification of tumour in intricate anatomical areas, resulting in more accurate surgical planning. A more precise delineation of nodal disease and metastasis will result in a more accurate and lesser surgical dissection, and consequent reduction in morbidity.

The PSMA-PET-CT will be compared with the standard-of-care imaging, FDG-PET-CT to evaluate utility of this approach. It is of note that FDG-PET CT has a high background FDG uptake normally seen in the brain and liver, and PSMA could potentially be a more favourable tracer if there is less background uptake.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥18 years of age
* Biopsy proven first and recurrent metastatic melanoma with palpable nodal disease who have undergone a staging FDG PET-CT scan as part of routine clinical care and are scheduled for surgery for resection of the primary site

Exclusion Criteria:

* Patients unable to give voluntary written informed consent to participate in this study
* Patients not willing to complete all the study assessments
* Patients who are females
* Patients who are taking androgen deprivation therapy (ADT) and other therapies targeting the androgen pathway, such as androgen receptor antagonists.
* Patients who have or have previously been diagnosed with prostate cancer
* Patients who have had Lu-177 PSMA therapy or barium studies within a period of 10 days prior to undergoing PSMA PET-CT scanning
* Patients not fluent in English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PSMA PET-CT detection of melanoma metastases | 1 Year
  The principal objective of the study is to investigate whether the diagnostic biomarker, prostate-specific membrane antigen (PSMA), can detect melanoma metastases using a PSMA PET/ CT.

SECONDARY OUTCOMES:
Compare FDG PET-CT & PSMA PET-CT | 1 Year
  1. To compare FDG PET-CT in identifying known metastasis with PSMA PET-CT
  2. To compare the radiological information obtained by FDG PET-CT and PSMA PET-CT

CONTACTS AND LOCATIONS:
Overall Officials: Myles Smith, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in Melanoma biomarkers. Data or samples shared will be coded, with no patient health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Analytic Code
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact (surgicalresearchteam@rmh.nhs.uk).